CLINICAL TRIAL: NCT06110156
Title: Population Health Approach to Optimizing and Deprescribing Medications in Older Adults
Brief Title: Population Health Approach to Optimizing Medications in Older Adults
Acronym: POP-MED
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Michelle Keller, Research Scientist I, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00002921; K01AG076865 (NIH)
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Medication Adverse Effects; Older Adults (65 Years and Older); Polypharmacy; Polypharmacy Patients; Deprescribing
Keywords: Older adults; Polypharmacy; Deprescribing
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Patient-tailored deprescribing assessment and intervention (MCI and Dementia diagnosis) (Experimental): Patients are identified for enrollment via a risk prediction model and enrolled in a pharmacist-led polypharmacy clinic. The pharmacist will conduct a comprehensive medication review, which will include: medication reconciliation, assessment of patient risk factors, identification of potentially inappropriate medications, identification of potential prescribing omissions, shared decision-making with the patient and/or caregiver, and confirmation of the results with the prescriber. Once the prescriber has approved the recommendations, the pharmacist will make the appropriate changes to the medication regimen, will provide tailored medication education and counseling and will follow-up with the patient at least once per month to assess side effects, adverse effects, and provide support. This arm specifically includes only patients with a diagnosis of Mild Cognitive Impairment (MCI) or Alzheimer's Disease and Related Dementias (ADRD) at enrollment.
  Interventions: Behavioral: Patient-tailored deprescribing assessment and intervention
- Usual care (MCI and Dementia diagnosis) (No Intervention): Patients in the comparator arm will see their primary care clinician as needed. This arm specifically includes patients with a diagnoses of Mild Cognitive Impairment (MCI) or Alzheimer's Disease and Related Dementias (ADRD) at enrollment.
- Patient-tailored deprescribing assessment and intervention (no MCI and Dementia diagnosis) (Experimental): Patients are identified for enrollment via a risk prediction model and enrolled in a pharmacist-led polypharmacy clinic. The pharmacist will conduct a comprehensive medication review, which will include: medication reconciliation, assessment of patient risk factors, identification of potentially inappropriate medications, identification of potential prescribing omissions, shared decision-making with the patient and/or caregiver, and confirmation of the results with the prescriber. Once the prescriber has approved the recommendations, the pharmacist will make the appropriate changes to the medication regimen, will provide tailored medication education and counseling and will follow-up with the patient at least once per month to assess side effects, adverse effects, and provide support. This arm specifically includes only patients with NO diagnosis of Mild Cognitive Impairment (MCI) or Alzheimer's Disease and Related Dementias (ADRD) at enrollment.
  Interventions: Behavioral: Patient-tailored deprescribing assessment and intervention
- Usual care (no MCI and Dementia diagnosis) (No Intervention): Patients in the comparator arm will see their primary care clinician as needed. This arm specifically includes patients with NO diagnoses of Mild Cognitive Impairment (MCI) or Alzheimer's Disease and Related Dementias (ADRD) at enrollment.

INTERVENTIONS:
Behavioral: Patient-tailored deprescribing assessment and intervention — Patients are identified for enrollment via a risk prediction model and enrolled in a pharmacist-led polypharmacy clinic. The pharmacist will conduct a comprehensive medication review, which will include: medication reconciliation, assessment of patient risk factors (clinical, socioeconomic), identification of potentially inappropriate medications, identification of potential prescribing omissions, shared decision-making with the patient and/or caregiver, and confirmation of the results of the comprehensive medication review with the primary care clinician. Once the primary care clinician has approved the recommendations, the pharmacist will make the appropriate changes to the medication regimen, will provide tailored medication education and counseling (including Motivational Interviewing) and will follow-up with the patient at least once per month via video visit or phone to assess side effects, adverse effects, and provide support.
  Arms: Patient-tailored deprescribing assessment and intervention (MCI and Dementia diagnosis); Patient-tailored deprescribing assessment and intervention (no MCI and Dementia diagnosis)

SUMMARY:
This randomized controlled pragmatic pilot study examines the feasibility and acceptability of a population health-based deprescribing intervention that leverages a polypharmacy risk prediction model. It includes four arms (2 intervention and 2 control arms) and uses a parallel arm study design.

DETAILED DESCRIPTION:
This pilot clinical trial will examine the feasibility and acceptability of a medication management intervention that uses risk stratification to identify older adults (including older adults with Mild Cognitive Impairment or Alzheimer's Disease and Related Dementias) at greatest risk for polypharmacy-related adverse events. The intervention will use a risk prediction model to identify potential study participants for inclusion and enroll them and their care partners into a polypharmacy clinic. The study will stratify patients by cognitive impairment status. The risk prediction model includes variables such as: age, sex, recent healthcare encounters, current and past medications, current and past lab tests, current and past diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be invited to enroll in the study if they are in the top decile of risk selected by a risk prediction model of polypharmacy-related adverse events. The risk prediction model includes variables such as: age, sex, recent healthcare encounters, current and past medications, current and past lab tests, current and past diagnoses.
* 65 years of age or older
* Have a primary care clinician within the Cedars-Sinai Health System who uses MyCSLink (electronic health record used by Cedars-Sinai).
* Part of a Cedars-Sinai Health System population health registry (e.g., enrolled in an Accountable Care Organization, Medicare Advantage plan, or Primary Care First program)
* Diagnosis of Mild Cognitive Impairment or Dementia at baseline (for one intervention group) on the problem list

Exclusion criteria include:

* Patients for whom there is an active substance use disorder (defined by a physician) and thus for whom the intervention may not be appropriate
* Patients with an organ transplant
* Visits with a Cedars-Sinai Medical Center pharmacist for a polypharmacy consult within the last 6 months
* Patients who previously indicated in the EHR that they wish to opt out of participating in research studies.
* Patients enrolled in CS360, a program for highly complex medical patients, who already receive polypharmacy services.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-11-24 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of all-cause hospitalizations | 12 months after enrollment
  Number of all-cause inpatient visits (including observation visits) 12 months after enrollment.

SECONDARY OUTCOMES:
Total number of medications | Baseline, 12 months
  Total number of medications on the medication list, including prescription medications, over-the-counter medications, vitamins, and supplements at 12 months.
Total number of potentially inappropriate medications | Baseline, 12 months
  Use of any potentially inappropriate medications, defined by the 2019 Beers Criteria Tables 2 and 7
Number of medications with a dose reduction >10% over 12 months | 12 months
  We will sum up the number of medications where the study participant has achieved at >10% dose reduction compared to baseline for each study participant at baseline and 12 months in both study arms.
Number of medications discontinued for 90 days or more which are re-prescribed | Baseline, 12 months
  We will sum up the number of medications where the study participant has had any re-prescription of medications which were discontinued for 90 days or more by 12 months in all study arms.
Number of times per day the patient is taking medications | Baseline, 12 months
  Each study participant will be coded on a continuous scale the number of times a day medications are taken based on the prescription instructions at baseline and 12 months in all study arms.
Number of potential prescribing omissions (PPOs) based on the STOPP/START criteria | 12 months
  Number of potential prescribing omissions (PPOs) based on the STOPP/START criteria
Number of drug-related problems | Baseline, 12 months
  We will compare the total number of drug-related problems (identified retrospectively by a pharmacist) at baseline and 12 months.
Number of potential pharmacy recommendations | Baseline, 12 months
  We will compare the total number of potential pharmacist recommendations (identified retrospectively by a pharmacist) at baseline and 12 months.
Change in risk prediction model score | 12 months
  Each study participant's information will be run through the risk prediction model at the end of the study to see if there is a meaningful change (10% or more change) in the risk prediction score from baseline to the end of the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Keller, PhD, MPH, Principal Investigator — University of Southern California
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No